CLINICAL TRIAL: NCT06334822
Title: Randomised Controlled Trial For Assessing The Effectiveness Of An Inclusive Heart Failure Monitoring And Tracking Solution In The UK.(HF-TRACK)
Brief Title: Randomised Controlled Trial for Assessing the Effectiveness of an Inclusive Heart Failure Monitoring and TRACKing Solution in the UK.
Acronym: HF-TRACK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heartfelt Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HFT-2024-01
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: peripheral oedema; Heart failure decompensation; Heart failure hospitalisation
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care; Surveys and Questionnaires; Dosage Forms

STUDY DESIGN:
Intervention Model Description: This 6-month study involves up to 210 patients using the Heartfelt device at home. It is a crossover trial with a 21-day break between two 69-day periods to prevent overlap effects. Patients will either receive standard care or standard care plus Heartfelt alerts. The Heartfelt group is further divided into three 23-day sub-studies to test different alert systems.
  Another 60 patients will have monthly measurements taken at the pharmacy without being part of the main randomisation.
Who Masked: Outcomes Assessor
Masking Description: Only outcomes assessors will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care + Heartfelt device (Experimental): In addition to standard care activities, participants have the Heartfelt device at home. During this arm, the device sends alerts and measurement data to the patient, carers and clinicians.
  Interventions: Device: Heartfelt Device installed; Other: Standard care; Other: Questionnaires; Device: Heartfelt device alerting system
- Standard care (control) (Active Comparator): In addition to standard care activities, participants have the Heartfelt device at home. During this arm, data is captured without sending health alerts or measurement data to the patient, carers and clinicians.
  Interventions: Device: Heartfelt Device installed; Other: Standard care; Other: Questionnaires
- Standard Care + Heartfelt device in pharmacy (Experimental): Participants will follow standard care advice, and have monthly measurements taken at the pharmacy using the Heartfelt device. The pharmacist will receive the measurements and alerts and be able to communicate this to the participant.
  Interventions: Other: Standard care; Other: Questionnaires; Device: Heartfelt Device in pharmacy

INTERVENTIONS:
Device: Heartfelt Device installed — Device installed in the patient's home and capturing foot volume data which are processed in the cloud.
  Other Names: Remote patient monitoring device
  Arms: Standard Care + Heartfelt device; Standard care (control)
Other: Standard care — Patients with heart failure are advised to weigh daily and to report weight increase to their clinician. They should also report changes in breathlessness, tiredness and other symptoms associated with heart failure decompensation.
  Other Names: Daily weighing, Breathlessness, Dizziness, Tiredness
Other: Questionnaires — Patients are presented with one or more optional questionnaires (some validated, some bespoke)
  Other Names: 5Q-5D, Bespoke Questionnaires
Device: Heartfelt Device in pharmacy — Device used monthly in the pharmacy, with the assistance of the pharmacist, and capturing foot volume data which are processed in the cloud.
  Other Names: Monitoring device used in phamarcy
  Arms: Standard Care + Heartfelt device in pharmacy
Device: Heartfelt device alerting system — The Heartfelt device sends alerts to the patients directly (audio-visual alert on the device, and app alerts), carers and/or medical professionals.
  Other Names: Remote patient monitoring device
  Arms: Standard Care + Heartfelt device

SUMMARY:
The objective of our research is to evaluate the effectiveness of an innovative medical device designed to measure foot and lower leg sizes in detecting early indications of deteriorating heart failure. This health condition frequently causes leg swelling and breathing difficulties due to fluid accumulation. Early detection of these symptoms is vital for effective management, potentially preventing the need for hospitalization.

Fluid retention in the lower legs and lungs, manifesting as swollen ankles and shortness of breath, is a common sign of progressing heart failure. Often, a slight increase in body weight is the first warning of fluid accumulation, occurring before noticeable swelling or breathing issues arise. Early identification of these fluid accumulation signs is critical for timely intervention, which can avert the necessity for hospital admittance. Patients are usually encouraged to monitor their weight, check for swelling in the ankles, observe their breathing, and consult with their healthcare provider or heart failure specialist at the first sign of these symptoms. In many cases, patients can report these symptoms in time for their healthcare team to adjust their treatment accordingly. Diuretics, or water pills, are often prescribed to help eliminate excess fluid, effectively preventing hospital admissions when used promptly.

The Heartfelt device may provide a useful solution for individuals who find it challenging to consistently monitor these indicators and their weight. It is designed to detect early warning signs seamlessly without imposing additional tasks on the patient's daily routine. The device, intended to complement rather than replace self-monitoring practices, is user-friendly and operates by scanning the feet for any size changes, positioned conveniently by the bedroom floor. This capability allows healthcare professionals to make informed decisions swiftly about patient care, potentially adjusting treatments to avoid further health complications. The device captures images of the feet only, ensuring privacy.

This study aims to ascertain the device's practical effectiveness in real-world scenarios, aiming to collect precise data to confirm its potential benefits for patients facing heart failure challenges.

DETAILED DESCRIPTION:
This study has been co-designed with existing and past users (patients and their carers) of the Heartfelt device who have in the past expressed an interest in sharing their opinion for future research.

It is a 6 months crossover randomised controlled trial designed to evaluate the effectiveness of the Heartfelt device, a remote patient monitoring system, in reducing the risk of hospitalisation for heart failure (HF) by monitoring peripheral oedema.

We will focus on patients with heart failure who have had at least one hospitalisation for heart failure associated with peripheral oedema in the last year, with stratified randomisation (for the RCT part) to avoid recent discharge effects in the early phases of data collection and focussing on patients considered at high-risk of poor long-term adherence to daily weights (the majority of patients with heart failure). [8-Fitzgerald].

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this trial, an individual must meet all of the following criteria:

* Provision of signed and dated informed consent form (e-consent via website or app is acceptable).
* Women or men, aged 18 years or older [No maximum age].
* Diagnosis of heart failure at least 3 months previously
* Receiving diuretics on a daily basis
* Peripheral oedema reported on at least one HF-related hospitalisation in the last 4 years (as documented in EPR).
* Hospitalised for HF OR on a Virtual Ward for HF OR has received IV diuretic treatment in the last 12 months, or treated with at least 80 mg furosemide (or equivalent) orally per day.
* For women of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 6 weeks after the end of the study.
* Is considered by the investigator to be non-adherent OR at high risk of HF hospital readmissions.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* bandages to lower limbs every day
* amputation of both feet
* regular wheelchair user inside their home
* bed-bound
* no fixed abode
* taking part in a conflicting evaluation/study that could confound the results of this evaluation and/or impact clinical interventions and participant outcomes
* Pregnancy or lack of contraceptive measures if of child-bearing potential†
* Inability to install the device (even with assistance) allowing at least 6 months of data capture by the end of the study.

Patients with severe aortic stenosis or awaiting a heart procedure or surgery

† This exclusion criterion has been requested by the insurance provider for clinical trial cover.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause Mortality Rate. | Through study completion, an average of 6 months
  This measure tracks the total number of participant deaths due to any cause during the study period. It is an essential indicator of overall participant survival and general safety of the treatment under investigation. This data is collected and verified through clinical records.
  Measure: The number of all-cause deaths documented in clinical records.
  Unit of Measure: Count of deaths.
Device-Related Complication Rate. | Through study completion, an average of 6 months
  This measure captures the frequency of complications associated with the medical device used in the study. It includes any adverse events or malfunctions linked to the device, providing insight into its safety and performance.
  Measure: The incidence of complications related to the medical device in use, as specified in Sections 8.1.4 and 8.1.5 of the study protocol.
  Unit of Measure: Count of complication events.
Heart Failure Hospitalisation Incidence. | Through study completion, an average of 6 months
  This metric quantifies the number of times participants are admitted to the hospital due to heart failure. The criteria for what constitutes a heart failure hospitalisation are based on the definition provided by Hicks KA in 2017, ensuring standardised and specific event classification.
  Measure: The frequency of hospital admissions specifically for heart failure, as defined by Hicks KA, 2017.
  Unit of Measure: Count of heart failure hospitalisation events.

SECONDARY OUTCOMES:
Cause of Death | Through study completion, an average of 6 months
  This records the cause of death classified as related to heart failure (HF) or not, as defined in Hicks KA, 2017.
  Measure: Cause of Death Unit of Measure: Date (YYYY-MM-DD)
Date of Death | Through study completion, an average of 6 months
  This records the date of death classified as related to heart failure (HF) or not, as defined in Hicks KA, 2017.
  Measure: Date of Death Unit of Measure: Categorical
Hospital Admission Duration | Through study completion, an average of 6 months
  Description:
  This measures the length of hospital stays, noting the admission and discharge dates.
  Measure: Length of Stay Unit of Measure: Days
Cause of Hospitalization | Through study completion, an average of 6 months
  This identifies the primary reason for hospitalization. Measure: Cause Hospitalization Category Unit of Measure: Categorical.
Hospitalisation Admission Route | Through study completion, an average of 6 months
  This identifies the route of admission during hospitalization events, such as ICU, CCU, or ward admission.
  Measure: Admission Route Unit of Measure: Categorical (ICU, CCU, Ward)
Loss of Independence | Through study completion, an average of 6 months
  This assesses instances where a patient becomes unable to live at home, necessitating care in a facility.
  Measure: Change in Living Arrangements Unit of Measure: Binary (Independent, Dependent)
Scheduling of Care Events | Through study completion, an average of 6 months
  This differentiates between scheduled and unscheduled care events. Measure: Nature of Scheduling Unit of Measure: Categorical (Scheduled, Unscheduled)
Setting of Care Events | Through study completion, an average of 6 months
  This categorizes care events as either inpatient or outpatient. Measure: Care Setting Unit of Measure: Categorical (Inpatient, Outpatient)
Date of Changes in HF Medication Post-Discharge | Through study completion, an average of 6 months
  This tracks the date of any change in heart failure medications after the patient returns home, excluding changes made during ward stays.
  Measure: Medication Adjustment Date Unit of Measure: Date (YYYY-MM-DD)
Changes in dosage of HF Medication Post-Discharge | Through study completion, an average of 6 months
  This tracks the change(s) in dosage in heart failure medications after the patient returns home, excluding changes made during ward stays.
  Measure: Medication Adjustment Dosage Unit of Measure: % change from previous dosage.
Comparison of Data Availability (number of days with data in a month): Heartfelt Device vs. Existing Remote Monitoring Devices | Through study completion, an average of 6 months
  This measures the variance in data availability, encompassing both device-generated and contemporaneous self-reported data.
  Measure: Degree of Variance Unit of Measure: Number of days per month with physiological measurements taken.
Timestamp of Health Alerts Generated by the Heartfelt Device | Through study completion, an average of 6 months
  This measures the date and time of health alerts generated by the Heartfelt device.
  Measure:
  Timestamp of Health Alerts
  Unit of Measure:
  Date and time
Frequency of Health Alerts Generated by the Heartfelt Device | Through study completion, an average of 6 months
  This measures the number of health alerts generated by the Heartfelt device over a specified period.
  Measure:
  Number of Health Alerts Unit of Measure: Count
Foot volume | Through study completion, an average of 6 months
  This reports the foot volume reported by the Heartfelt device. Measure: Foot and lower leg volume Unit of Measure: mL
Weight | Through study completion, an average of 6 months
  This measures the patient's weight Measure: patient weight Unit of Measure: Kg
Peripheral oedema grading | Through study completion, an average of 6 months
  This reports the Peripheral oedema grading reported by the Heartfelt device. Measure: Peripheral oedema grading Heartfelt scale [0-None / 1-Mild (includes ankle, but no higher) / 2-Moderate (Above the ankle, up to and including the knee)/ 4-Severe (Above the knee)]

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - The Ridings Medical Group, Brough, East Riding of Yorkshire
  - Dr R Raut & Partnership (General Practice), Hull, East Riding of Yorkshire
  - Croydon Health Services NHS Trust, Croydon, London
  - Barking, Havering and Redbridge University Hospitals NHS Trust, London, London
  - West Suffolk NHS Foundation Trust, Bury St Edmunds, Suffolk
  - Modality East Surrey Medical Practice, Horley, Surrey
  - Modality Partnership Airedale, Wharfedale & Craven:, Keighley, West Yorkshire
  - Pillsorted Ltd, Cambridge
  - Sutton Manor Pharma Services, Hull

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.

REFERENCES:
- [Result] Hicks KA, Mahaffey KW, Mehran R, Nissen SE, Wiviott SD, Dunn B, Solomon SD, Marler JR, Teerlink JR, Farb A, Morrow DA, Targum SL, Sila CA, Hai MTT, Jaff MR, Joffe HV, Cutlip DE, Desai AS, Lewis EF, Gibson CM, Landray MJ, Lincoff AM, White CJ, Brooks SS, Rosenfield K, Domanski MJ, Lansky AJ, McMurray JJV, Tcheng JE, Steinhubl SR, Burton P, Mauri L, O'Connor CM, Pfeffer MA, Hung HMJ, Stockbridge NL, Chaitman BR, Temple RJ; Standardized Data Collection for Cardiovascular Trials Initiative (SCTI). 2017 Cardiovascular and Stroke Endpoint Definitions for Clinical Trials. Circulation. 2018 Feb 27;137(9):961-972. doi: 10.1161/CIRCULATIONAHA.117.033502. PMID 29483172